CLINICAL TRIAL: NCT01730313
Title: Treatment of Nodding Syndrome - A Randomized Blinded Placebo-Controlled Crossover Trial of Oral Pyridoxine and Conventional Anti-Epileptic Therapy, in Northern Uganda - 2012
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Did not get approval from the collaborating partners in-country
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Ministry of Health, Uganda (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDC-CGH-6318
Record Dates: First submitted 2012-11-09; First posted 2012-11-21 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Nodding Syndrome
Keywords: Nodding syndrome
MeSH Terms: conditions — Nodding Syndrome | interventions — Pyridoxine; Vitamin B 6; Valproic Acid; Phenytoin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Pyridoxine (B6) (Experimental): Oral pyridoxine, 30- 50 mg/kg/day in one daily dose (powder form)for a period of four weeks followed by cross-over to Phenytoin arm for another four weeks
  Interventions: Drug: Pyridoxine; Drug: Phenytoin
- Phenytoin (Experimental): Phenytoin Oral, 5 mg/kg/day in two equally divided doses(powder form)for a period of four weeks and then cross-over to Pyridoxine arm for another four weeks
  Interventions: Drug: Pyridoxine; Drug: Phenytoin
- Sodium Valproate (Experimental): Sodium valproate oral, 10 - 15 mg/kg/day once daily powder form)for a period of four weeks and then cross-over to placebo arm for another four weeks
  Interventions: Drug: Sodium Valproate; Drug: Placebo
- Placebo (Placebo Comparator): Placebo will consist of an inert substance (e.g., gelatin) with an appearance similar to medication in similar dosage as the study arms for a period of 4 weeks and subsequent cross-over to Sodium Valproate arm
  Interventions: Drug: Sodium Valproate; Drug: Placebo

INTERVENTIONS:
Drug: Pyridoxine
  Other Names: Vitamin B6
  Arms: Phenytoin; Pyridoxine (B6)
Drug: Sodium Valproate
  Arms: Placebo; Sodium Valproate
Drug: Phenytoin
  Arms: Phenytoin; Pyridoxine (B6)
Drug: Placebo
  Arms: Placebo; Sodium Valproate

SUMMARY:
Nodding Syndrome (NS) is a novel form of epilepsy seen predominantly among children aged 5-15 years and characterized by head nodding, progressively worsening seizures, and cognitive impairment. To date, the cause of NS remains unclear. A recent assessment by the Uganda Ministry of Health (MOH), World Health Organization (WHO), and US CDC conducted in Kitgum District in northern Uganda documented that the nodding episodes themselves resulted from atonic seizures, and that the children also exhibit multiple different seizure types, both clinically and electrographically. The investigation also found that there was significantly greater sero-positivity for onchocerciasis among children with NS compared with control children, and demonstrated low serum concentrations of vitamin B6 (pyridoxine) among both cases and controls. Vitamin B6 is involved in neurotransmission and has been an effective treatment of seizures for certain rare type of epileptic syndrome. Children with nodding syndrome in Kitgum have been episodically treated with multivitamins, ivermectin, and anti-epileptic medications including phenobarbital, phenytoin, carbamazepine, and valproate, but the possible beneficial or harmful effects of any of these medications for nodding syndrome has not been systematically assessed, and reports from parents and guardians about apparent effectiveness are varied.

The investigators propose a randomized blinded four group clinical trial with crossover design to study the effect and response to therapeutic doses of oral pyridoxine (vitamin B6) and treatment with currently used conventional anti-epileptics including phenytoin and sodium valproate, among children with nodding syndrome.

DETAILED DESCRIPTION:
Nodding Syndrome (NS) is described as an epileptic seizure disorder and has been documented in various geographic areas of sub-Saharan Africa. Jilek et al, 1962, first described several children with attacks of 'nodding head' in Mahenge, a region in southern Tanzania (1,2,3). A missionary doctor described children in southern Sudan in the mid-1990s, where it was first noted in the Lui and Amadi villages of East Mundri county and the Lui region of western Equatoria; a medical NGO then reported the condition to WHO in 1997. An estimated 300 cases were reported in 2003 from this region (4, 5). Winkler et al., using data from Tanzania provided a clinical classification of seizures, semiology and socio-cultural aspects suggesting it was a syndrome (referred to as "head-nodding syndrome") and a form of epilepsy (6, 7). In 2008 and 2009, reports of an illness consistent with NS were reported in Kitgum and Pader districts, northern Uganda. Kaiser et al, in 2009, referred to the phenomenon of head nodding as possibly constituting a feature of an epileptic syndrome caused by O. volvulus (8).

Descriptions of the features of NS appear similar between reports (Appendix A). Nodding is frequently described as occurring in response to some stimulus, frequently being the presence of food or exposure to cold (4, 5, 6, 7). The nodding consists of repetitive bobbing or nodding of the head, sometimes associated with loss of muscle tone in the trunk and upper extremities (6, 7). Consciousness may or may not be impaired during the nodding episodes. The syndrome has been described to be progressive, with gradual neurological deterioration and development of additional seizure types, developmental regression, cognitive decline, and sometimes reportedly resulting in serious injuries or death both due to accidental falls into fires or wells during seizure episodes. Treatment with conventional antiepileptic medications has anecdotally been reported to result in some symptomatic improvement of both nodding and other seizure types. Health workers in southern Sudan report that children who start treatment early and on regular basis have seizures less frequently (9).

The cause of NS is unknown. Various factors and exposures have been postulated to cause NS, including exposure to munitions, prior history of measles infection, consumption of baboon meat and sorghum, and others. Two recent case-control investigations, one conducted among children with NS in Uganda during 2009 - 2010 and another conducted in S. Sudan in 2011 (below) have not supported these associations. One risk factor that appears to consistently demonstrate an association with NS is evidence of infection, past or present, with the microfilarial parasite Onchocerca volvulus, or a similar microfilarial parasite that is serologically cross-reactive with Onchocerca. O. volvulus is transmitted by black flies. Clinical manifestation of onchocerciasis is mainly ocular, with resultant vision loss due to inflammatory keratitis ("River Blindness"). A significant association of NS with detection of O. volvulus microfilariae in skin snips was observed in a case-control investigation in Sudan in 2001 - 2002, and in an assessment in Tanzania (84% of 62 children with NS had microfilariae or O. volvulus nucleic acid in skin snips). Various studies and reviews have identified an association between onchocerciasis and epilepsy in general (5, 10, 11, 12, 13, 14, 15, 16, 17, 44, 46). A high prevalence of seizure disorders in onchocerciasis endemic areas was noted in Western Equatoria in 1946.

In the WHO investigations conducted in southern Sudan in late 2001, skin snip positivity and higher microfilaria loads of O. volvulus were found in children with NS when compared to children without the condition, consistent with similar observations of a possible association between seizures and onchocerciasis from other studies (5, 10, 11, 12, 13, 14, 15, 16, 17, 44, 46). These, and subsequent investigations in 2002 by WHO could not identify any environmental pollutants, chemical agents or food toxins, nor several infectious agents, as possible causes for the seizures. EEG among 31 children assessed showed progressive epileptic encephalopathy.

In December 2009, a team from the US Centers for Disease Control and Prevention (CDC) assisted the Uganda Ministry of Health and the WHO in the investigation of the occurrence of NS in Kitgum / Pader regions of northern Uganda. A total of 51 cases with reported NS, and 93 household or friend controls were identified for the case control investigation and additionally, 23 subjects with reported NS were enrolled in a case series that underwent thorough medical and neurological assessments.

Unpublished data from the assessment demonstrated that NS is a seizure disorder, and that the nodding episodes are due to atonic seizures resulting in loss of tone associated with changes on electroencephalography (EEG) including multiple other clinical and subclinical seizure types. The surveillance data showed that the prevalence of NS in parts of Kitgum region is many-fold higher than what would be expected for comparable forms of epilepsy, based upon data from North America and Europe.

In the case-control investigation, while skin snip positivity for the presence of O. volvulus microfilariae was not associated with NS cases, seropositivity for antibodies to O. volvulus was, with 95% of cases positive for onchocerciasis serology compared with 54% of controls (p=0.03). The investigation also showed low serum vitamin B6 (pyridoxine) levels (<20) among the population of children between the ages of 5 and 15 in the region as a whole, both cases and controls. Deficiencies in vitamin A, selenium, and zinc, among both cases and controls were also noted.

The Ministry of Health, Government of Southern Sudan (MoH-GoSS), further investigated for NS in the Witto internally displaced persons (IDP) camp in Witto Payam in western Equatoria in September 2010. A total of 96 cases were registered, most aged between 5-20 years (highest in the age group 10-15 years). Head nodding, tonic-clonic partial seizures with secondary generalization and generalized seizures were reported. Based on the past two investigations, and available data, it was concluded that NS is a form of epilepsy with causes remaining obscure (9).

In May and June of 2011, a team from the CDC assisted the South Sudan Ministry of Health and the WHO with an investigation of NS in Western Equatoria State in South Sudan. A total of 38 case-control pairs matched by age- and village- were identified for the case control investigation and separately, 25 subjects with reported NS were enrolled in a case series and underwent thorough medical and neurological evaluations (17). The findings from this investigation were consistent with the unpublished findings from investigations in Uganda in 2009-10, with the cause of Nodding syndrome continuing to remain unknown.

Currently, parents and caregivers of children with NS report that children respond to locally available anti-epileptic drugs (AEDs) differently; some reporting that there is a response and others not. These locally available AEDs include carbamazepine, phenytoin, phenobarbitone, and valproate. However, this information is anecdotal and it remains unclear whether children receive medications on a regular basis, what doses are administered or adhered to, or whether they achieve therapeutic levels of AEDs. The investigators therefore additionally propose two AED treatment arms with conventional anti-epileptic therapy including sodium valproate and phenytoin, in order to validate the reported response to conventional anti-epileptic drugs.

Based on investigations done so far, children with NS appear to suffer from multiple clinical and electrographic seizure types, including generalized tonic-clonic, partial complex, atypical absence, and atonic seizures. Seizures are classified as partial generalized, and unclassified based on the clinical features and associated electroencephalographic findings (Appendix Y). There are many causes for seizures, including infectious, metabolic, drugs, genetic, nutritional, endocrinal, and trauma. In some cases, an etiology is not known, and the seizures are referred to as idiopathic or cryptogenic. Currently, because an etiology for NS has not been identified, the children suffer from multiple different seizure types, and many children demonstrate cognitive impairment, NS could be considered a form of cryptogenic epileptic encephalopathy. This is important because such epilepsies can be very difficult to control with standard AEDs, and in some cases, may be exacerbated with certain AEDs (e.g., carbamazepine) (18, 19, 20, 21, 22). Thus, a formal assessment of the effects of AEDs on children with NS is important.

The finding of low pyridoxine levels among children assessed, in the population of Kitgum District as well as in the children assessed in Western Equatoria in South Sudan is notable, in the light of a condition known as pyridoxine-dependent seizures (PDS) and pyridoxine-responsive seizures. Hunt et al, (1954) first described pyridoxine dependent seizures (PDS) (23) with an autosomal recessive inheritance. PDS is due to defective binding of pyridoxine to its apoenzyme, glutamate decarboxylase, which catalyzes the conversion of glutamic acid, a critical nutrient, into gamma-aminobutyric acid (GABA), an inhibitory central nervous system neurotransmitter. The resultant reduced levels of GABA lower the seizure threshold, leading to intractable seizures (24, 25,26, 27, appendix Z).

PDS commonly manifests among infants as intractable seizures, generally beginning within hours of birth. Classically multiple types of clinical and electrographic seizures are described among individuals with PDS (24, 28, 29, 30). Prolonged seizures and recurrent episodes of status epilepticus are typical, also reported are recurrent self-limited events including partial seizures, generalized seizures, atonic seizures, myoclonic events, and infantile spasms (27, 30, 31).

Commonly seen in neonates and infants, atypical presentations are known to occur with seizure onset later in childhood including report in a child of 6 years (26, 27, 32, 33, 34).

PDS is a diagnostic consideration in such instances among infants when the seizures are intractable and may not be controlled with conventional anticonvulsants but that respond both clinically and electrographically to pharmacologic doses of pyridoxine (27, 35).

A trial of therapeutic doses of B6 (administration of 100 mg or more of pyridoxine) is indicated in infants / children with intractable seizures unresponsive to standard anti-epileptic drug (AED) treatment (24, 25, 26, 35, 36, 37, 38). Intravenous or intramuscular administration is recommended in infants with ongoing seizures or status epilepticus, in order to achieve immediate resolution of seizures and clinical seizures generally cease over several minutes to hours (29). If responsive, oral maintenance dose of 2-500mg/day PO (15-18mg/kg/day optimally and sometimes as high as 680mg initially and 200 mg/day subsequently) has to be followed indefinitely (33, 35). Clinical seizures generally cease over several minutes to hours. Recommended daily allowance (RDA) for pyridoxine is 0.5 mg for infants and 2.0 mg for adults or 50-100 mg of pyridoxine per day (38, 39, 40) with dosage adjustment for age, intercurrent illnesses and to allow greatest intellectual performance but not exceeding 500 mg/day (27, 28, 36, 38, 41). The chance to identify specificity is lost if pyridoxine is given together with or after, many anticonvulsant drugs (27). Daily supplementation with pharmacologic doses of pyridoxine is the accepted treatment for this disorder.

The seizures as reported to occur among children with NS appear to share several features with PDS, namely multiple seizure types. However, NS does not represent PDS in its typical form; any relationship between NS and pyridoxine deficiency is only suspected in light of the presence of the deficiency in the population. However, unpublished findings from two investigations undertaken separately in Uganda (2010) and South Sudan (2011) show that deficiency of B6 has been noticed among this population of children (both cases and controls) raises the possibility of a contributory role of B6 deficiency in NS. Since the entire population, including both children with and without NS, appears to be pyridoxine-deficient, the illness cannot be attributed to B6 deficiency alone; however, the possibility that low B6 levels may be a contributory factor remains and therefore a treatment trial with pyridoxine is proposed because PDS is a therapeutic diagnostic consideration in such settings. Because the seizures in children with NS appear to have a gradual onset, and are intermittent with significant interictal periods, intravenous administration of pyridoxine is not necessary and oral supplementation will be most appropriate. B6 treatment is safe. There are few reports of significant side effects of B6 treatment. Apnea, lethargy and hypotonia among infants soon after starting B6 have been reported (3 out of 5 infants by Mikati, et al), but these are rare (29).

Since the diagnosis of PDS is based upon a response to the therapeutic intervention and requires a trial of the treatment, and such replacement may provide a safe, efficacious treatment for PDS, we propose to assess the possible efficacy of B6 supplementation for NS in the form of oral pyridoxine treatment to evaluate the response and efficacy on the cessation or reduction of seizures. Dosing for pyridoxine is 30 - 50 mg/kg/day in a single daily dose.

In summary, there appears to be growing data that NS is a seizure disorder and some of the various current treatment approaches have focused on use of antiepileptic medications. For most Ugandan children with this disorder, the current standard is no treatment or episodic treatment with multivitamins and/or antiepileptic medications, which are typically administered by psychiatric nurses with no or limited physician oversight. Information about the effectiveness of this treatment approach is based on anecdotal reports, and there are no reliable systematically collected data about dosage or frequency of medication use. In addition to the lack of scientific data on the effectiveness of these treatment approaches, there are important questions that need to be addressed regarding possible adverse effects of use of antiepileptic medications in children with NS. Anecdotal reports from caregivers and local treating physicians suggest that NS seizures appear to respond variably to locally available anti-epileptic drugs; however, for the reasons outlined above, this has not been clearly demonstrated. In addition, several aspects of treatment remain undetermined including, whether children are given medications on a regular basis, are given appropriate doses of antiepileptic drugs per weight, or are achieving therapeutic doses of drug.

In addition, it is not clear whether the children with NS are obtaining clinical benefit or are being harmed from AED treatment. Given the knowledge on the nature of the seizure types seen in NS, it is possible that NS will be difficult to manage with conventional AED approaches. In fact, certain antiepileptic medications may in some cases paradoxically exacerbate certain seizure conditions (18, 19, 20, 21, 22). Such exacerbation is particularly true in epileptic encephalopathies. For children with cryptogenic generalized epileptic disorders, the AED sodium valproate (valproic acid) has been found to be often effective, has fewer side effects than many other AEDs, and is considered the drug of choice (42). Valproic acid is currently listed as a recommended AED by WHO. The investigators therefore propose a simultaneous assessment of pyridoxine, valproic acid, as well as an AED that is currently being utilized in the community for children with NS (phenytoin) and compare them with response if any to a placebo controlled intervention group.

ELIGIBILITY:
Inclusion Criteria: All children identified at clinic level and/or community level in the study region will be eligible to enter into the study if they meet the following inclusion criteria after completing the screening form (Appendix H):

1. Clinical head nodding episodes with or without other types of seizure activity with a frequency of at least 1 per day (7 episodes per week). [The seizures must be frequent enough so that a change/decrease in that frequency is measurable.] Children will be stratified into those with high frequency or observed nodding (with 3 or more episodes daily), and lower frequency events (more than one but fewer than 3 episodes per day reported).
2. Plan to remain in the study area/region for at least two months from the time of entry
3. Are attended by a care giver who is/are able to understand and give informed consent
4. Are at least 5 years old at the time of entry into the study and not more than 17 years

Exclusion Criteria: Children will not be eligible for registration (or will be excluded from the trial if already registered) if they are determined to meet any of the following exclusion criteria when screened initially or at the time of entry into study:

1. Have a history of allergic reaction to any anti-epileptic medications
2. Have severe acute malnutrition diagnosed based on anthropometric measurements
3. Have known or suspected condition in which anti-epileptic medications or pyridoxine treatment is contraindicated
4. Because both phenytoin and valproate have been associated with birth defects and adverse events on the developing fetus, pregnancy will be ruled out before inclusion of females reaching menarche. Pregnant females will not be included in the study.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change in the frequency of observed head nodding and other seizure activity from baseline (which is the frequency at week 1) | 1 week, 5 weeks, 7 weeks, 12 weeks
  Change (Reduction) in frequency of observed head nodding or other seizure activity episodes among children with NS

CONTACTS AND LOCATIONS:
Overall Officials: Scott Dowell, MD, Principal Investigator — Centers for Disease Control and Prevention; JAMES SEJVAR, MD, Principal Investigator — Centers for Disease Control and Prevention; SUDHIR BUNGA, MD, Principal Investigator — Centers for Disease Control and Prevention; RICHARD IDRO, MD, Principal Investigator — Ministry of Health, Uganda
Locations (1):
- Kitgum Nodding Syndrome Treatment Center, Kitgum General Hospital, Kitgum, Uganda